CLINICAL TRIAL: NCT01396746
Title: Cardiovascular Function in Sub Maximal Exercise and Performance in Three Daily Activity Tests in Persons With Post Stroke Conditions
Brief Title: Cardiovascular Function in Sub Maximal Exercise and Performance in Three Daily Activity Tests After Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: Zinman College of Physical Education and Sports Sciences (Other); Israel Sport Center for the Disabled (Other)
Responsible Party: Dr. Avraham Katz, Israel Sport Center for the Disabled
Other Study IDs: 54-2011
Record Dates: First submitted 2011-06-28; First posted 2011-07-19 (Estimated); Last update posted 2011-07-19 (Estimated); Status verified 2011-07

CONDITIONS: Stroke; Hemiplegia
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- People with Post Stroke Conditions: (a) having acquired stroke at least 1 year before testing. (b) Chronic weakness and/or spasticity of the affected side. (c) Independent stair-climbers (with hand-rail). (d) With cognitive level sufficient to comprehend instructions. (e) age range between 40-69. (f) Use of walking aid is permitted as long as the participant is able to walk on a treadmill with hand-rail. (g) No heart failure or other medical conditions that preclude participation in the study.

SUMMARY:
The purpose of this study is to explore the relationship between cardiovascular function of persons with post stroke conditions and their performance in three field tests. This is a validation study, aiming to determine during which of two activities VO2 measurements better express the functional restrictions caused by stroke, And to find out whether the Total Heart Beat Index can be used in the case of stroke survivors for the prediction of mechanical efficiency when measured during stair-climbing and of energy cost during treadmill walking.

The hypothesis is that Stair Climbing (STC) is a more suitable form of exercise capacity testing compared to Treadmill Walk (TMW) since it potentially requires a greater amount of external work, and therefore will show stronger correlation with functional tests demonstrating the same ability, whereas TMW does not utilize the movement capability of participants to the fullest.

Another hypothesis is that cardiac response to the exertion can be used as a predictor of those measures during these exertions in the post stroke population.

ELIGIBILITY:
Inclusion Criteria:

* Having acquired stroke at least 1 year before testing
* Chronic weakness and/or spasticity of the affected side
* Independent stair-climbers (with hand-rail)
* Received medical clearance from a physician
* With cognitive level sufficient to comprehend instructions
* Participants' age will range between 40-69
* Use of walking aid is permitted as long as the participant is able to walk on a treadmill with hand-rail.

Exclusion Criteria:

* Unable to understand instructions
* Unable to ambulate
* Severe aphasia
* Heart failure or other medical conditions that preclude participation in the study.

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are recruited in community centers designated for Disabled populations. They are leading a physically active life style, usually facilitated by an assistant.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-06

PRIMARY OUTCOMES:
Exercise VO2 | 60 days
Exercise HR | 60 days
Mechanical efficiency | 60 days
Time for-Up-and-go (TUG) Test | 60 days
Time for 10 m walk test | 60 days
Distance for 6 min walk test | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Yeshayahu Hutzler, Dr., Study Chair — The Wingate institute for physical education and sports; Avraham Katz, MD, Principal Investigator — Israel Sport Center for the Disabled; Galia Modai, Study Director — The Wingate Institute for Physical Education and Sports
Locations (1):
- Israel Sport Center for the Disabled, Ramat Gan, Israel

REFERENCES:
- [Background] Andriacchi TP, Andersson GB, Fermier RW, Stern D, Galante JO. A study of lower-limb mechanics during stair-climbing. J Bone Joint Surg Am. 1980 Jul;62(5):749-57. PMID 7391098
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Bar-Haim S, Belokopytov M, Harries N, Loeppky JA, Kaplanski J. Prediction of mechanical efficiency from heart rate during stair-climbing in children with cerebral palsy. Gait Posture. 2008 Apr;27(3):512-7. doi: 10.1016/j.gaitpost.2007.06.006. Epub 2007 Aug 8. PMID 17689964
- [Background] Berg KO, Wood-Dauphinee SL, Williams JI, Maki B. Measuring balance in the elderly: validation of an instrument. Can J Public Health. 1992 Jul-Aug;83 Suppl 2:S7-11. PMID 1468055
- [Background] Blum L, Korner-Bitensky N. Usefulness of the Berg Balance Scale in stroke rehabilitation: a systematic review. Phys Ther. 2008 May;88(5):559-66. doi: 10.2522/ptj.20070205. Epub 2008 Feb 21. PMID 18292215
- [Background] Bowen TR, Lennon N, Castagno P, Miller F, Richards J. Variability of energy-consumption measures in children with cerebral palsy. J Pediatr Orthop. 1998 Nov-Dec;18(6):738-42. PMID 9821128
- [Background] Carvalho C, Willen C, Sunnerhagen KS. Relationship between walking function and 1-legged bicycling test in subjects in the later stage post-stroke. J Rehabil Med. 2008 Oct;40(9):721-6. doi: 10.2340/16501977-0242. PMID 18843423
- [Background] Chen G, Patten C, Kothari DH, Zajac FE. Gait differences between individuals with post-stroke hemiparesis and non-disabled controls at matched speeds. Gait Posture. 2005 Aug;22(1):51-6. doi: 10.1016/j.gaitpost.2004.06.009. PMID 15996592
- [Background] Crenna P. Spasticity and 'spastic' gait in children with cerebral palsy. Neurosci Biobehav Rev. 1998 Jul;22(4):571-8. doi: 10.1016/s0149-7634(97)00046-8. PMID 9595571
- [Background] Crompton S, Khemlani M, Batty J, Ada L, Dean C, Katrak P. Practical issues in retraining walking in severely disabled patients using treadmill and harness support systems. Aust J Physiother. 2001;47(3):211-3. doi: 10.1016/s0004-9514(14)60268-3. No abstract available. PMID 11552877
- [Background] da Cunha-Filho IT, Henson H, Wankadia S, Protas EJ. Reliability of measures of gait performance and oxygen consumption with stroke survivors. J Rehabil Res Dev. 2003 Jan-Feb;40(1):19-25. PMID 15150717
- [Background] de Oliveira CB, de Medeiros IR, Frota NA, Greters ME, Conforto AB. Balance control in hemiparetic stroke patients: main tools for evaluation. J Rehabil Res Dev. 2008;45(8):1215-26. PMID 19235121
- [Background] Detrembleur C, Dierick F, Stoquart G, Chantraine F, Lejeune T. Energy cost, mechanical work, and efficiency of hemiparetic walking. Gait Posture. 2003 Oct;18(2):47-55. doi: 10.1016/s0966-6362(02)00193-5. PMID 14654207
- [Background] Donnan GA, Davis SM. Breaking the 3 h barrier for treatment of acute ischaemic stroke. Lancet Neurol. 2008 Nov;7(11):981-2. doi: 10.1016/S1474-4422(08)70230-8. No abstract available. PMID 18940690
- [Background] Duncan PW, Sullivan KJ, Behrman AL, Azen SP, Wu SS, Nadeau SE, Dobkin BH, Rose DK, Tilson JK; LEAPS Investigative Team. Protocol for the Locomotor Experience Applied Post-stroke (LEAPS) trial: a randomized controlled trial. BMC Neurol. 2007 Nov 8;7:39. doi: 10.1186/1471-2377-7-39. PMID 17996052
- [Background] Fulk GD, Echternach JL, Nof L, O'Sullivan S. Clinometric properties of the six-minute walk test in individuals undergoing rehabilitation poststroke. Physiother Theory Pract. 2008 May-Jun;24(3):195-204. doi: 10.1080/09593980701588284. PMID 18569856
- [Background] Gordon NF, Duncan JJ. Effect of beta-blockers on exercise physiology: implications for exercise training. Med Sci Sports Exerc. 1991 Jun;23(6):668-76. PMID 1679517
- [Background] Gordon NF, Gulanick M, Costa F, Fletcher G, Franklin BA, Roth EJ, Shephard T; American Heart Association Council on Clinical Cardiology, Subcommittee on Exercise, Cardiac Rehabilitation, and Prevention; the Council on Cardiovascular Nursing; the Council on Nutrition, Physical Activity, and Metabolism; and the Stroke Council. Physical activity and exercise recommendations for stroke survivors: an American Heart Association scientific statement from the Council on Clinical Cardiology, Subcommittee on Exercise, Cardiac Rehabilitation, and Prevention; the Council on Cardiovascular Nursing; the Council on Nutrition, Physical Activity, and Metabolism; and the Stroke Council. Circulation. 2004 Apr 27;109(16):2031-41. doi: 10.1161/01.CIR.0000126280.65777.A4. No abstract available. PMID 15117863
- [Background] Hood VL, Granat MH, Maxwell DJ, Hasler JP. A new method of using heart rate to represent energy expenditure: the Total Heart Beat Index. Arch Phys Med Rehabil. 2002 Sep;83(9):1266-73. doi: 10.1053/apmr.2002.34598. PMID 12235607
- [Background] Kelly-Hayes M, Robertson JT, Broderick JP, Duncan PW, Hershey LA, Roth EJ, Thies WH, Trombly CA. The American Heart Association Stroke Outcome Classification. Stroke. 1998 Jun;29(6):1274-80. doi: 10.1161/01.str.29.6.1274. No abstract available. PMID 9626308
- [Background] Kollen B, van de Port I, Lindeman E, Twisk J, Kwakkel G. Predicting improvement in gait after stroke: a longitudinal prospective study. Stroke. 2005 Dec;36(12):2676-80. doi: 10.1161/01.STR.0000190839.29234.50. Epub 2005 Nov 10. PMID 16282540
- [Background] Lamontagne A, Stephenson JL, Fung J. Physiological evaluation of gait disturbances post stroke. Clin Neurophysiol. 2007 Apr;118(4):717-29. doi: 10.1016/j.clinph.2006.12.013. Epub 2007 Feb 16. PMID 17307395
- [Background] Lord SE, Rochester L. Measurement of community ambulation after stroke: current status and future developments. Stroke. 2005 Jul;36(7):1457-61. doi: 10.1161/01.STR.0000170698.20376.2e. Epub 2005 Jun 9. PMID 15947265
- [Background] Mathias S, Nayak US, Isaacs B. Balance in elderly patients: the "get-up and go" test. Arch Phys Med Rehabil. 1986 Jun;67(6):387-9. PMID 3487300
- [Background] Meyring S, Diehl RR, Milani TL, Hennig EM, Berlit P. Dynamic plantar pressure distribution measurements in hemiparetic patients. Clin Biomech (Bristol). 1997 Jan;12(1):60-65. doi: 10.1016/s0268-0033(96)00050-2. PMID 11415673
- [Background] IJzerman MJ, Baardman G, van 't Hof MA, Boom HB, Hermens HJ, Veltink PH. Validity and reproducibility of crutch force and heart rate measurements to assess energy expenditure of paraplegic gait. Arch Phys Med Rehabil. 1999 Sep;80(9):1017-23. doi: 10.1016/s0003-9993(99)90054-0. PMID 10489002
- [Background] Nakamura R, Handa T, Watanabe S, Morohashi I. Walking cycle after stroke. Tohoku J Exp Med. 1988 Mar;154(3):241-4. doi: 10.1620/tjem.154.241. PMID 3376101
- [Background] Neptune RR, Sasaki K, Kautz SA. The effect of walking speed on muscle function and mechanical energetics. Gait Posture. 2008 Jul;28(1):135-43. doi: 10.1016/j.gaitpost.2007.11.004. Epub 2007 Dec 26. PMID 18158246
- [Background] Pang MY, Eng JJ, Dawson AS. Relationship between ambulatory capacity and cardiorespiratory fitness in chronic stroke: influence of stroke-specific impairments. Chest. 2005 Feb;127(2):495-501. doi: 10.1378/chest.127.2.495. PMID 15705987
- [Background] Perron M, Malouin F, Moffet H. Assessing advanced locomotor recovery after total hip arthroplasty with the timed stair test. Clin Rehabil. 2003 Nov;17(7):780-6. doi: 10.1191/0269215503cr696oa. PMID 14606746
- [Background] Perry J. The mechanics of walking in hemiplegia. Clin Orthop Relat Res. 1969 Mar-Apr;63:23-31. No abstract available. PMID 5769371
- [Background] Pizzi A, Carlucci G, Falsini C, Lunghi F, Verdesca S, Grippo A. Gait in hemiplegia: evaluation of clinical features with the Wisconsin Gait Scale. J Rehabil Med. 2007 Mar;39(2):170-4. doi: 10.2340/16501977-0026. PMID 17351701
- [Background] Pohl M, Mehrholz J, Ritschel C, Ruckriem S. Speed-dependent treadmill training in ambulatory hemiparetic stroke patients: a randomized controlled trial. Stroke. 2002 Feb;33(2):553-8. doi: 10.1161/hs0202.102365. PMID 11823669
- [Background] Pohl PS, Duncan PW, Perera S, Liu W, Lai SM, Studenski S, Long J. Influence of stroke-related impairments on performance in 6-minute walk test. J Rehabil Res Dev. 2002 Jul-Aug;39(4):439-44. PMID 17638141
- [Background] Raine AE, Pickering TG. Cardiovascular and sympathetic response to exercise after long-term beta-adrenergic blockade. Br Med J. 1977 Jul 9;2(6079):90-2. doi: 10.1136/bmj.2.6079.90. PMID 17451
- [Background] RALSTON HJ. Energy-speed relation and optimal speed during level walking. Int Z Angew Physiol. 1958;17(4):277-83. doi: 10.1007/BF00698754. No abstract available. PMID 13610523
- [Background] Sims NR, Muyderman H. Mitochondria, oxidative metabolism and cell death in stroke. Biochim Biophys Acta. 2010 Jan;1802(1):80-91. doi: 10.1016/j.bbadis.2009.09.003. Epub 2009 Sep 12. PMID 19751827
- [Background] Tang A, Sibley KM, Bayley MT, McIlroy WE, Brooks D. Do functional walk tests reflect cardiorespiratory fitness in sub-acute stroke? J Neuroeng Rehabil. 2006 Sep 29;3:23. doi: 10.1186/1743-0003-3-23. PMID 17010203
- [Background] Teixeira-Salmela LF, Nadeau S, Mcbride I, Olney SJ. Effects of muscle strengthening and physical conditioning training on temporal, kinematic and kinetic variables during gait in chronic stroke survivors. J Rehabil Med. 2001 Mar;33(2):53-60. doi: 10.1080/165019701750098867. PMID 11474950
- [Background] van de Port IG, Wood-Dauphinee S, Lindeman E, Kwakkel G. Effects of exercise training programs on walking competency after stroke: a systematic review. Am J Phys Med Rehabil. 2007 Nov;86(11):935-51. doi: 10.1097/PHM.0b013e31802ee464. PMID 17303962
- [Background] Vanhees L, Fagard R, Amery A. Influence of beta adrenergic blockade on effects of physical training in patients with ischaemic heart disease. Br Heart J. 1982 Jul;48(1):33-8. doi: 10.1136/hrt.48.1.33. PMID 6123335
- [Background] von Schroeder HP, Coutts RD, Lyden PD, Billings E Jr, Nickel VL. Gait parameters following stroke: a practical assessment. J Rehabil Res Dev. 1995 Feb;32(1):25-31. PMID 7760264
- [Background] Waters RL, Mulroy S. The energy expenditure of normal and pathologic gait. Gait Posture. 1999 Jul;9(3):207-31. doi: 10.1016/s0966-6362(99)00009-0. PMID 10575082
- [Background] Werner C, Von Frankenberg S, Treig T, Konrad M, Hesse S. Treadmill training with partial body weight support and an electromechanical gait trainer for restoration of gait in subacute stroke patients: a randomized crossover study. Stroke. 2002 Dec;33(12):2895-901. doi: 10.1161/01.str.0000035734.61539.f6. PMID 12468788
- [Background] Wevers L, van de Port I, Vermue M, Mead G, Kwakkel G. Effects of task-oriented circuit class training on walking competency after stroke: a systematic review. Stroke. 2009 Jul;40(7):2450-9. doi: 10.1161/STROKEAHA.108.541946. Epub 2009 May 21. PMID 19461035
- [Background] Zamparo P, Francescato MP, De Luca G, Lovati L, di Prampero PE. The energy cost of level walking in patients with hemiplegia. Scand J Med Sci Sports. 1995 Dec;5(6):348-52. doi: 10.1111/j.1600-0838.1995.tb00057.x. PMID 8775719